CLINICAL TRIAL: NCT03141099
Title: Blood Pressure and Oxygenation Targets in Post-resuscitation Care, a Randomized Clinical Trial
Brief Title: Blood Pressure and OXygenation Targets After OHCA
Acronym: BOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jesper Kjaergaard (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Sponsor-Investigator, Jesper Kjaergaard, MD, Ph.d., DMSc., Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-16033436
Record Dates: First submitted 2017-04-30; First posted 2017-05-04 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Out-of-Hospital Cardiac Arrest; Blood Pressure; Hemodynamic Instability
Keywords: OHCA; Hemodynamic; TTM; post-rescusitation care; Blood pressure targets; Oxygenation targets
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized trial in 2*2 factorial design allocating comatose OHCA patients to one of two target blood pressures (double blind) and restrictive vs. liberal oxygenation (open label) during ICU stay with blinded outcome evaluation.
  Sample size: 800 patients. Patient will be allocated 1:1; for all interventions, no interaction with regards to outcome is expected.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Target blood pressure will be blinded by offsetting the blood pressure measurering module.
  The oxygenation- and fever control interventions will be open label. Further life-sustaining treatment will be delivered according to standard procedures and withdrawal of active intensive care will be at the discretion of the treating physicians, but must be delayed for at least 108 hours post ROSC. The steering group and the management group will be blinded to the type of intervention during the entire trial period, when handling the trial database.
  Follow-up at 30 days (phone call) and 90 days (meeting) will be performed by personnel unaware of the allocation group, treatment complications at the ICU, if they occurred or specialized neurological rehabilitation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low normal MAP and low normal PaO2 (Active Comparator): MAP 63 mmHg and PaO2 9-10 kPa during targeted temperature management (36 hours) after OHCA.
  Interventions: Other: Low normal MAP; Other: Low normal PaO2.
- High normal MAP and low normal PaO2 (Active Comparator): MAP 77 mmHg and PaO2 9-10 kPa during targeted temperature management (36 hours) after OHCA.
  Interventions: Other: High normal MAP; Other: Low normal PaO2.
- Low normal MAP and high normal PaO2 (Active Comparator): MAP 63 mmHg and PaO2 13-14 kPa during targeted temperature management (36 hours) after OHCA.
  Interventions: Other: Low normal MAP; Other: High normal PaO2
- High normal MAP and high normal PaO2 (Active Comparator): MAP 77 mmHg and PaO2 13-14 kPa during targeted temperature management (36 hours) after OHCA.
  Interventions: Other: High normal MAP; Other: Low normal PaO2.

INTERVENTIONS:
Other: Low normal MAP — The patients are randomized to recieve a Phillips M1006B blood pressure measuring module, offset by +10 %. All patients will target a MAP of 70, but due to the offset module, the patients will target an actual blood pressure of 63 mmHg.
  Other Names: Mean arterial blood pressure at 63 mmHg.
  Arms: Low normal MAP and high normal PaO2; Low normal MAP and low normal PaO2
Other: High normal MAP — The patients are randomized to recieve a Phillips M1006B blood pressure measuring module, offset by -10 %. All patients will target a MAP of 70, but due to the offset module, the patients will target an actual blood pressure of 77mmHg.
  Other Names: Mean arterial blood pressure at 77 mmHg .
  Arms: High normal MAP and high normal PaO2; High normal MAP and low normal PaO2
Other: Low normal PaO2. — The patients are randomized to a PaO2 target of 9-10 kPa (open-label).
  Other Names: PaO2 at 9-10 kPa.
  Arms: High normal MAP and high normal PaO2; High normal MAP and low normal PaO2; Low normal MAP and low normal PaO2
Other: High normal PaO2 — The patients are randomized to a PaO2 target of 13-14 kPa (open-label).
  Other Names: PaO2 at 13-14 kPa.
  Arms: Low normal MAP and high normal PaO2

SUMMARY:
This study compares two blood pressure targets and two oxygenation targets in the post-resuscitation care of comatose out-of-hospital cardiac arrets patients. Using a novel method the blood pressure-intervention is double-blinded. The oxygenation-intervention is open-label. As a subordinate study, the patients will be randomized 1:1 to active fever-control with an automated feedback temperature control-device for 36 or 72 hours following return of spontaneous circulation.

DETAILED DESCRIPTION:
In comatose patients resuscitated from out of hospital cardiac arrest (OHCA), neurological injuries remain the leading cause of death. The in-hospital mortality is reported at 30-50%, and the total mortality, although improved substantially over the last decade, remain to be significant, in most countries at up to 90%. An adequate blood pressure must be maintained in the post-cardiac arrest patient i order to optimize neurological recovery and avoid further brain injury. Blood pressure targets in post-resuscitation guidelines are based on limited clinical evidence. Furthermore registry and clinical data suggest a u-shaped relationship of outcome with levels of oxygen supplementation. Blinded, randomized, clinical trials addressing specific blood pressure- or oxygenation-targets during the post-resuscitation care, have not been performed.

The current trial addresses strategies for neuroprotection using a 2-by-2 design of two different target blood pressure levels and two different oxygenation levels.

Intervention:

* 'Low-normal MAP' (appoximately 63 mmHg) vs. 'high-normal MAP' (approximately 77 mmHg) (double blind intervention) and
* Low-normal oxygenation (9-10 kPa) vs. high-normal oxygenation (13-14) kPa (open label).
* As a subordinate study, the patients will be randomized 1:1 to active fever-control with an automated feedback temperature control device for 72 hours or to 36 hours following return of spontaneous circulation.

Design: National collaborative, randomized clinical trial randomizing 800 comatose out-of-hospital cardiac arrest patients undergoing targeted temperature management (TTM) to the specified interventions.

The investigators have planned the following sub-studies:

Sub-study 1: Devopment and validation af a method for double blinded allocation to different blood pressure targets.

Hypothesis: It is possible to develop a method for double blinded allocation of patients to different blood pressure targets in clinical trials.

Sub-study 2: Assessment of different blood pressure targets and relation to renal function during TTM.

Hypothesis: Different blood presure goals will affect biomarkes of renal function after cardiac arrest.

Sub-study 3: To investigate the hemodynamic profil in relation to different blood pressure targets after cardiac arrest.

Hypothesis: Blood pressure and vassopressor-doses are related to hemodynamic parameters, such as systemic vaskular resistence index and cardiac index.

Sub-study 4: To investigate the hemodynamic profil in relation to different oxygenation targets after cardiac arrest.

Hypothesis: Lower oxygenation targets are related to higher pulmonary vascular resistance.

Sub-study 5: The prognostic value of automated videobased assessment of pupillary dilatation and reaction to light. Derivation and validation of relevant cut-off for introducing pupillomtry as part of the prognostication

INTERIM ANALYSIS There will be an independent DSMC arranging an independent statistician to conduct primarily a blinded interim analysis at time points of their choosing. The DSMC will be able to request unblinding of data coordinated by the data managing agency. An interim analysis is planned after inclusion of 200 and 400 patients.

For the BP intervention, a blinded interim analysis of vasorepressor need and recorded blood pressures is planned after 50 patients, to monitor blinding of treatment allocation and that a clinically relevant blood pressure separation between groups is achieved. Vasopressor needs in terms of vasopressor need in a variance component model is expected to differ. New sites will be monitored for these factors after inclusion of 50 patients.

EARLY STOPPING CRITERIA After an interim analysis the DSMC may suggest to the steering committee that the trial should be stopped early. No specific criteria to guide the DSMB will be put forward.

ACCOUNTABILITY PROCEDURE FOR MISSING DATA/POPULATION FOR ANALYSIS Trial sites will be asked to complete all CRFs and other forms if missing data is found in the electronic database. Missing data will be reported in the publications. More than 5% missing data will result in multiple imputation with the creation of 5-10 imputed datasets to be analysed separately and the aggregated into one estimate of intervention effect on the primary and secondary outcomes. Analyses will be performed according to the modified intention to treat principle with patients lost to follow up included in the denominator.

SUBGROUP ANALYSIS AND DESIGN VARIABLES Subgroups will be analysed according to pre-defined design variables: over or under median age, shockable rhythm, gender, the presence of shock at admission, diagnosed AMI and time from arrest to ROSC. Difference in intervention effect estimates according to subgroup will be declared exclusively based on a statistically significant test of interaction.

DIRECT ACCESS TO SOURCE DATA/DOCUMENTATION The principal investigator and the site investigators will permit monitoring, audits, review of ethical committees and regulatory authorities direct access to source data and documentation, blinded to treatment allocation.

DATA HANDLING AND RECORD KEEPING Individual patient data will be handled as ordinary chart records and will be kept according to the legislation (e.g. data protection agencies) of the countries of each health system. The study database will be stored for 15 years and anonymised if requested by the relevant authorities.

Danish legislation regarding the respect for patients physical and mental integrity and rights will be respected, Approval for storing data relevant to the trial, including potentially sensitive information has been approved by the relevant authorities.

QUALITY CONTROL AND QUALITY ASSURANCE A monitoring plan will be published before start of the trial. The monitoring will include: inclusion and absence of exclusion criteria, consent obtained in all patients.

All trial sites will be provided with sufficient information to participate in the trial. The site investigator will be responsible for that all relevant data is entered into the electronic CRFs. The CRFs will be constructed in order to assure data quality with predefined values and ranges on all data entries.

STATISTICAL METHODS The combined primary outcome will be reported as proportional hazard of experiencing one of two endpoints (death or poor neurological status at hospital discharge), differences tested with a log rank test. Other proportions are expected to be normally distributed; therefore a t-test is applied. Survival analyses are performed using proportional hazard models, survival is adjusted for site.

Furthermore pre-specified analysis of interaction for design variables: sex, age (median), time to ROSC (median), shockable rhythm, STEMI, pre-existing hypertension, pre-existing chronic obstructive pulmonary disease.

SIGNIFICANCE A two-sided significance level of 0.05 will be applied to all endpoints. No adjustment for the factorial design is made, as no interaction is expected.

SAMPLE SIZE ESTIMATION Sample size estimation is based on blinded BP target allocation and on the assumption that no interaction of the two interventions exist.

The combined primary outcome is time to death or hospital discharge in a state of CPC 3 or 4. The investigators are planning a study with 400 subjects in each group, an accrual interval of 48 months, and additional follow-up after the accrual interval of 3 months. Prior data indicate the 6 months mortality is 33% overall. Assuming a mortality of 28% in the superior group compared to 38% in the inferior groups the investigators will need to include 732 patients in total or 846 patients in total to achieve a power of 0.8 and 0.9 respectively. The Type I error probability associated with this test of the null hypothesis that the experimental and control survival curves are equal is 0.05.

Loss of final measurement is expected but from the experience from previous trial the number of missing follow-up assessments is small (<5%) and will not result in an increase of the number of patients needed.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. OHCA of presumed cardiac cause
3. Sustained ROSC
4. Unconsciousness (GCS <8) (patients not able to obey verbal commands) after sustained ROSC

Exclusion Criteria:

1. Conscious patients (obeying verbal commands)
2. Females of childbearing potential (unless a negative HCG test can rule out pregnancy within the inclusion window)
3. In-hospital cardiac arrest (IHCA)
4. OHCA of presumed non-cardiac cause, e.g. after trauma or dissection/rupture of major artery OR Cardiac arrest caused by initial hypoxia (i.e. drowning, suffocation, hanging).
5. Known bleeding diathesis (medically induced coagulopathy (e.g. warfarin, NOAC, clopidogrel) does not exclude the patient).
6. Suspected or confirmed acute intracranial bleeding
7. Suspected or confirmed acute stroke
8. Unwitnessed asystole
9. Known limitations in therapy and Do Not Resuscitate-order
10. Known disease making 180 days survival unlikely
11. Known pre-arrest CPC 3 or 4
12. >4 hours (240 minutes) from ROSC to screening
13. Systolic blood pressure <80 mm Hg in spite of fluid loading/vasopressor and/or inotropic medication/intra-aortic balloon pump/axial flow device
14. Temperature on admission <30°C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 802 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
All-cause mortality or severe anoxic brain injury | 3 months after OHCA.
  Death from any cause or discharge from hospital in Cerebral Performance Category 3 or 4

SECONDARY OUTCOMES:
Renal replacement therapy | 3 months
  Time to Renal replacement therapy.
Time to death | 180 days
  Time to death
Neuron-Specific Enolase | 48 hours
  Neuron-Specific Enolase level at 48 hours
MOCA-score | 3 months
  Assesed at three months (lowest score allocated to patients not available for follow-up).
Modified Ranking Scale | 3 months
  Modified Ranking Scale.
NT-pro-BNP | 3 months
  NT-pro-BNP at three months (Highest value allocated to patients not available for follow-up).
eGFR | 3 months
  Last available measurement of eGFR with 3 month of follow-up
LVEF | 3 months
  Last available measurement of LVEF with 3 month of follow-up
Vasopressor use | First week after cardiac arrest
  Daily cumulated vasopressor requirement in the first week of the ICU stay.
Renal function | 96 hours
  Assesed by creatinine-clearence at 48 and 96 hours after OHCA.

OTHER OUTCOMES:
Vital status at 180 days post cardiac arrest | 180 days post cardiac arrest
  Vital status at 180 days post cardiac arrest
CPC category at 180 days post cardiac arrest | 180 days post cardiac arrest
  CPC category at 180 days post cardiac arrest

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Kjaergaard, Md, DMSc, Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Department of Cardiology, Copenhagen University Hospital, Rigshospitalet, Copenhagen, København Ø
  - Depart med Cardiothoracic Intensive Care, Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No
Will be shared by a case-by-case agreement

REFERENCES:
- [Derived] Meyer MAS, Beske RP, Molstrom S, Grand J, Obling LER, Wiberg S, Borregaard B, Schneekloth S, Kaad SG, Christensen PM, Christoffersen C, Frikke-Schmidt R, Schmidt H, Moller JE, Kjaergaard J, Hassager C. Neurofilament light chain for prognostication after cardiac arrest-first steps towards validation. Crit Care. 2025 Aug 6;29(1):348. doi: 10.1186/s13054-025-05579-1. PMID 40770665
- [Derived] Linde L, Beske RP, Meyer MAS, Molstrom S, Grand J, Helgestad OKL, Ravn HB, Schmidt H, Kjaergaard J, Hassager C, Moller JE. Hemodynamic Characteristics and Prognostic Implication of Modified Society for Cardiovascular Angiography and Interventions Shock Classification in Comatose Patients With Out-of-Hospital Cardiac Arrest. J Am Heart Assoc. 2025 Jan 7;14(1):e036659. doi: 10.1161/JAHA.124.036659. Epub 2024 Dec 20. PMID 39704227
- [Derived] Grand J, Granholm A, Wiberg S, Schmidt H, Moller JE, Molstrom S, Meyer MAS, Josiassen J, Beske RP, Dahl JS, Obling LER, Frydland M, Borregaard B, Lind Jorgensen V, Hartvig Thomsen J, Aalbaek Madsen S, Nyholm B, Hassager C, Kjaergaard J. Lower vs. higher blood pressure targets during intensive care of comatose patients resuscitated from out-of-hospital cardiac arrest-a Bayesian analysis of the BOX trial. Eur Heart J Acute Cardiovasc Care. 2025 Jan 31;14(1):14-23. doi: 10.1093/ehjacc/zuae142. PMID 39658315
- [Derived] Nyholm B, Grand J, Obling LER, Hassager C, Moller JE, Schmidt H, Othman MH, Kondziella D, Horn J, Kjaergaard J. Validating quantitative pupillometry thresholds for neuroprognostication after out-of-hospital cardiac arrest. A predefined substudy of the Blood Pressure and Oxygenations Targets After Cardiac Arrest (BOX)-trial. Intensive Care Med. 2024 Sep;50(9):1484-1495. doi: 10.1007/s00134-024-07574-6. Epub 2024 Aug 20. PMID 39162825
- [Derived] Grand J, Hassager C, Schmidt H, Molstrom S, Nyholm B, Obling LER, Meyer MAS, Illum E, Josiassen J, Beske RP, Hoigaard Frederiksen H, Dahl JS, Moller JE, Kjaergaard J. Impact of Blood Pressure Targets in Patients With Heart Failure Undergoing Postresuscitation Care: A Subgroup Analysis From a Randomized Controlled Trial. Circ Heart Fail. 2024 Jun;17(6):e011437. doi: 10.1161/CIRCHEARTFAILURE.123.011437. Epub 2024 Jun 7. PMID 38847097
- [Derived] Jeppesen KK, Rasmussen SB, Kjaergaard J, Schmidt H, Molstrom S, Beske RP, Grand J, Ravn HB, Winther-Jensen M, Meyer MAS, Hassager C, Moller JE. Acute kidney injury after out-of-hospital cardiac arrest. Crit Care. 2024 May 18;28(1):169. doi: 10.1186/s13054-024-04936-w. PMID 38762578
- [Derived] Meyer MAS, Hassager C, Molstrom S, Borregaard B, Grand J, Nyholm B, Obling LER, Beske RP, Meyer ASP, Bekker-Jensen D, Winther-Jensen M, Jorgensen VL, Schmidt H, Moller JE, Kjaergaard J. Combined effects of targeted blood pressure, oxygenation, and duration of device-based fever prevention after out-of-hospital cardiac arrest on 1-year survival: post hoc analysis of a randomized controlled trial. Crit Care. 2024 Jan 12;28(1):20. doi: 10.1186/s13054-023-04794-y. PMID 38216985
- [Derived] Grand J, Hassager C, Schmidt H, Molstrom S, Nyholm B, Hoigaard HF, Dahl JS, Meyer M, Beske RP, Obling L, Kjaergaard J, Moller JE. Serial assessments of cardiac output and mixed venous oxygen saturation in comatose patients after out-of-hospital cardiac arrest. Crit Care. 2023 Oct 27;27(1):410. doi: 10.1186/s13054-023-04704-2. PMID 37891623
- [Derived] Rasmussen SB, Jeppesen KK, Kjaergaard J, Hassager C, Schmidt H, Molstrom S, Beske RP, Grand J, Ravn HB, Winther-Jensen M, Meyer MAS, Moller JE. Blood Pressure and Oxygen Targets on Kidney Injury After Cardiac Arrest. Circulation. 2023 Dec 5;148(23):1860-1869. doi: 10.1161/CIRCULATIONAHA.123.066012. Epub 2023 Oct 4. PMID 37791480
- [Derived] Nyholm B, Grand J, Obling LER, Hassager C, Moller JE, Schmidt H, Othman MH, Kondziella D, Kjaergaard J. Quantitative pupillometry for neuroprognostication in comatose post-cardiac arrest patients: A protocol for a predefined sub-study of the Blood pressure and Oxygenations Targets after Out-of-Hospital Cardiac Arrest (BOX)-trial. Resusc Plus. 2023 Sep 26;16:100475. doi: 10.1016/j.resplu.2023.100475. eCollection 2023 Dec. PMID 37779885
- [Derived] Hassager C, Schmidt H, Moller JE, Grand J, Molstrom S, Beske RP, Boesgaard S, Borregaard B, Bekker-Jensen D, Dahl JS, Frydland MS, Hofsten DE, Isse YA, Josiassen J, Lind Jorgensen VR, Kondziella D, Lindholm MG, Moser E, Nyholm BC, Obling LER, Sarkisian L, Sondergaard FT, Thomsen JH, Thune JJ, Veno S, Wiberg SC, Winther-Jensen M, Meyer MAS, Kjaergaard J. Duration of Device-Based Fever Prevention after Cardiac Arrest. N Engl J Med. 2023 Mar 9;388(10):888-897. doi: 10.1056/NEJMoa2212528. Epub 2022 Nov 6. PMID 36342119
- [Derived] Schmidt H, Kjaergaard J, Hassager C, Molstrom S, Grand J, Borregaard B, Roelsgaard Obling LE, Veno S, Sarkisian L, Mamaev D, Jensen LO, Nyholm B, Hofsten DE, Josiassen J, Thomsen JH, Thune JJ, Lindholm MG, Stengaard Meyer MA, Winther-Jensen M, Sorensen M, Frydland M, Beske RP, Frikke-Schmidt R, Wiberg S, Boesgaard S, Lind Jorgensen V, Moller JE. Oxygen Targets in Comatose Survivors of Cardiac Arrest. N Engl J Med. 2022 Oct 20;387(16):1467-1476. doi: 10.1056/NEJMoa2208686. Epub 2022 Aug 27. PMID 36027567
- [Derived] Kjaergaard J, Moller JE, Schmidt H, Grand J, Molstrom S, Borregaard B, Veno S, Sarkisian L, Mamaev D, Jensen LO, Nyholm B, Hofsten DE, Josiassen J, Thomsen JH, Thune JJ, Obling LER, Lindholm MG, Frydland M, Meyer MAS, Winther-Jensen M, Beske RP, Frikke-Schmidt R, Wiberg S, Boesgaard S, Madsen SA, Jorgensen VL, Hassager C. Blood-Pressure Targets in Comatose Survivors of Cardiac Arrest. N Engl J Med. 2022 Oct 20;387(16):1456-1466. doi: 10.1056/NEJMoa2208687. Epub 2022 Aug 27. PMID 36027564
- [Derived] Kjaergaard J, Schmidt H, Moller JE, Hassager C. The "Blood pressure and oxygenation targets in post resuscitation care, a randomized clinical trial": design and statistical analysis plan. Trials. 2022 Feb 24;23(1):177. doi: 10.1186/s13063-022-06101-6. PMID 35209951
- [Derived] Grand J, Hassager C, Schmidt H, Moller JE, Molstrom S, Nyholm B, Kjaergaard J. Hemodynamic evaluation by serial right heart catheterizations after cardiac arrest; protocol of a sub-study from the Blood Pressure and Oxygenation Targets after Out-of-Hospital Cardiac Arrest-trial (BOX). Resusc Plus. 2021 Dec 10;8:100188. doi: 10.1016/j.resplu.2021.100188. eCollection 2021 Dec. PMID 34950913